CLINICAL TRIAL: NCT07061561
Title: Objective Evaluation of Cough Effort in Tracheotomized Patients (LOST Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0095_KINESITHERAPIE_LOST
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Tracheostomy; Cough; Weaning; Respiratory Function Tests; Diaphragm
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group - Cough Effort Measurement and Follow-Up (Other)
  Interventions: Device: Peak Expiratory Flow Measurement Using Peak Flow Meter and Lorio Device

INTERVENTIONS:
Device: Peak Expiratory Flow Measurement Using Peak Flow Meter and Lorio Device — This intervention involves the use of two respiratory measurement devices to assess cough strength in tracheotomized patients: the traditional Peak Flow meter, which measures peak expiratory flow (PEF), and the Lorio device, a novel tool designed for respiratory rehabilitation with customizable training exercises. Measurements are taken at multiple time points before and after decannulation to compare accuracy, reproducibility, and patient usability.

SUMMARY:
This study aims to evaluate how well tracheotomized patients can cough before and after their tracheostomy tube is removed. Cough strength is measured using two different tools-Peak Flow and Lorio. Researchers want to find out if the cough measurement taken before removing the tube can help predict how effective the patient's cough will be afterward. The study will also explore factors that might influence cough strength and compare the usefulness of the two tools. Additionally, it will assess how patients feel about using these devices and the role of diaphragm ultrasound in predicting cough effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Hospitalized in post-intensive care rehabilitation unit (SRPR) or intensive care unit (ICU)
* Tracheotomized during the weaning process
* Medical prescription for physiotherapy assessment
* Medical prescription for speech therapy assessment

Exclusion Criteria:

* Patients who have undergone total laryngectomy
* Patients with severe swallowing disorders
* Patients with cognitive impairments incompatible with understanding instructions
* Patients under medical decision to stop active treatments
* Patients who refuse to participate or refuse to sign informed consent
* Patients under guardianship or curatorship
* Patients not affiliated with a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of Peak Expiratory Flow (PEF) Measured Before Decannulation for PEF After Decannulation in Tracheotomized Patients. | From pre-decannulation measurement (up to 7 days before) to 72 hours after decannulation.